CLINICAL TRIAL: NCT07013617
Title: Effect Of Hamstring Stretch On Clinical Outcomes In Patellofemoral Pain Syndrome
Brief Title: Effect of Specific Versus General Hamstring Stretch on Clinical Outcomes in Patellofemoral Pain Syndrome (PFPS)
Acronym: PFPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amna Ibrahim Mahmoud Mohammed Shemila, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005812
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hamstring Shortness; Patellofemoral Pain Syndrome; Hamstring Flexibility; Patellofemoral Pain (PFPS)
Keywords: patellofemoral pain syndrome; PFPS; hamstring flexibility; active knee extension test; medial hamstring; lateral hamstring; specific hamstring stretch; Muscle Energy Technique; TENS; Visual Analogue Scale; Hand Held Dynamometer (HHD); Kujala Score
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (general hamstring stretch group) (Active Comparator): * General hamstring Muscle energy technique (MET)
  * TENS 20 min
  * Hip/knee strengthening program
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation Device; Other: Strength exercises for lower limb; Other: Hamstring Stretch Muscle Energy Technique(MET) (General )
- Arm B (medial hamstring stretch) (Active Comparator): * Medial hamstring MET
  * TENS 20 min
  * Hip/knee strengthening program
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation Device; Other: Strength exercises for lower limb; Other: Medial Hamstring Muscle energy technique(MET) stretch
- Arm C (lateral hamstring stretch) (Active Comparator): * Lateral hamstring MET
  * TENS 20 min
  * Hip/knee strengthening program
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation Device; Other: Strength exercises for lower limb; Other: Lateral hamstring Muscle Energy Technique(MET)Stretch

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation Device — Each participant will receive 20 minutes of TENS, Electrodes will be positioned around the patella with a 5 - 7 cm distance in between, The TENS settings include a continuous asymmetric biphasic square-pulse wave, a pulse width of 120 microseconds, and a pulse rate of 180 Hz.
  Other Names: TENS
Other: Strength exercises for lower limb — Each participant will receive progressive strengthening program targeting the hip and knee, begin with 3 sets of 10 repetitions and progress to 3 sets of 20 repetitions.
Other: Hamstring Stretch Muscle Energy Technique(MET) (General ) — The participant will be supine and the leg will be taken into hip flexion until a tightness is felt then patient will be asked to push down with his lower leg and hold the contraction for 10 seconds then relax for 2 to 3 seconds then the therapist will take the patient's leg into further flexion for 30 seconds this will be repeated for 3 times each session .
  Other Names: Non-Specific hamstring stretch MET
  Arms: Arm A (general hamstring stretch group)
Other: Medial Hamstring Muscle energy technique(MET) stretch — The Participant will be supine' then the therapist will take his leg in flexion, abduction and external rotation at the same time until he feels tightness then he will ask the patient to push his leg down and in or toward him and hold the contraction for 10 seconds then relax for 2 to 3 seconds then therapist will take the patient's leg in more abduction 'external rotation and flexion for 30 seconds, this will be repeated for 3 times each session
  Other Names: specific medial hamstring MET stretch
  Arms: Arm B (medial hamstring stretch)
Other: Lateral hamstring Muscle Energy Technique(MET)Stretch — The Participant will be supine' then the therapist will take his leg in flexion, adduction and internal rotation at the same time until he feels a tightness then he will ask the patient to push his leg down and out or away from him him and hold the contraction for 10 seconds then relax for 2 to 3 seconds then therapist will take the patient's leg in more adduction 'internal rotation and flexion for 30 seconds, this will be repeated for 3 times each session
  Other Names: Specific lateral hamstring MET stretch
  Arms: Arm C (lateral hamstring stretch)

SUMMARY:
This randomized, Single-blind, parallel-group trial will compare the effects of three hamstring stretching interventions-general hamstring Muscle Energy Technique (MET), medial hamstring MET, and lateral hamstring MET-each combined with standardized TENS and progressive hip/knee strengthening, on hamstring flexibility (knee-extension ROM), anterior knee pain (Arabic Kujala score), pain intensity visual analogue scale (VAS), and lower-limb strength (hand-held dynamometer) in adults with patellofemoral pain syndrome (PFPS).

DETAILED DESCRIPTION:
Patients with chronic PFPS will be randomized (1:1:1) into:

General MET group: standard non-specific hamstring MET stretch

Medial MET group: targeted medial-hamstring MET stretch

Lateral MET group: targeted lateral-hamstring MET stretch

All groups receive:

TENS: 20 min asymmetric biphasic square-pulse, 120 μs pulse width, 180 Hz, electrodes around patella (5-7 cm apart)

Strengthening: 3×/week for 4 weeks; hip/knee exercises, start 3×10 reps → 3×20, progress with weights or resistance bands.

Outcomes are measured pre-intervention and at 4 weeks. Analysis by mixed-design MANOVA (α < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Anterior or retropatellar knee pain lasting at least three months
* Pain reproduced by at least two functional tasks: squatting, kneeling, prolonged sitting, stair climbing, hopping or running
* Pain intensity of ≥3 on a Visual Analog Scale
* positive active knee extension test (inability to achieve greater than 160° of knee extension with the hip at 90° of flexion)
* Body mass index (BMI) < 30 Kg/m² and > 18Kg/m²

Exclusion Criteria:

* Previous knee surgery
* History of knee pathologies, such as meniscal injury' ligament injury, or knee osteoarthritis
* Psychological, cardiovascular' or neurological disorders
* Dizziness or fainting while doing exercises, pregnancy, or any contraindications to exercise
* Physical therapy treatment in the last 3 months

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
hamstring flexibility (knee extension range of motion ) | 4 weeks
  measuring knee extension range of motion(hamstring flexibility) by active knee extension test using kinovea software
Arabic Kujala Anterior knee pain score | 4 weeks
  Arabic Kujala Anterior knee pain score is used to measure pain and functional activities in anterior knee pain patients consisting of 13 questions, the Patient will be asked to mark the most suitable answer for him. Each answer has points up to 5 or 10, and the total score is 100.
  The higher the score, the better for the patient.

SECONDARY OUTCOMES:
pain intensity by visual analogue scale (VAS) | 4 weeks
  from 0 to 10 centimeter line patient will detect on it the usual pain felt and the worst pain during the day
lower limb strength using handheld dynamometer | 4 weeks
  using handheld dynamometer to assessment the strength of hip abductor, extensors, external rotators and knee extensors

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zahra Rojhani-Shirazi, Mohamad Reza Salimifard, Fatemeh Barzintaj. Comparison of the effects of static stretching and muscle energy technique on Hamstring flexibility, pain, and function in athletes with patellofemoral pain. J Adv Pharm Edu Res 2021;11(S1):33-38.
- [Background] Lopes HS, Waiteman MC, Priore LB, Glaviano NR, Bazett-Jones DM, Briani RV, Azevedo FM. There is more to the knee joint than just the quadriceps: A systematic review with meta-analysis and evidence gap map of hamstring strength, flexibility, and morphology in individuals with gradual-onset knee disorders. J Sport Health Sci. 2024 Jul;13(4):521-536. doi: 10.1016/j.jshs.2023.08.004. Epub 2023 Sep 3. PMID 37669706
- [Background] Wallis JA, Roddy L, Bottrell J, Parslow S, Taylor NF. A Systematic Review of Clinical Practice Guidelines for Physical Therapist Management of Patellofemoral Pain. Phys Ther. 2021 Mar 3;101(3):pzab021. doi: 10.1093/ptj/pzab021. PMID 33533400
- [Background] Hamdan M, Haddad B, Isleem U, Hamad A, Hussein L, Shawareb Y, Hadidi F, Alryalat SA, Samarah O, Khanfar A, Alzoubi B. Validation of the Arabic version of the Kujala patellofemoral pain scoring system. J Orthop Sci. 2019 Mar;24(2):290-293. doi: 10.1016/j.jos.2018.09.008. Epub 2018 Oct 10. PMID 30316659
- [Background] John Gibbons. (2022). Muscle energy techniques: a practical guide for physical therapists / JOHN GIBBONS (second edition). Lotus publishing / North Atlantic book
- [Background] Puig-Divi A, Escalona-Marfil C, Padulles-Riu JM, Busquets A, Padulles-Chando X, Marcos-Ruiz D. Validity and reliability of the Kinovea program in obtaining angles and distances using coordinates in 4 perspectives. PLoS One. 2019 Jun 5;14(6):e0216448. doi: 10.1371/journal.pone.0216448. eCollection 2019. PMID 31166989
- [Background] Hott A, Brox JI, Pripp AH, Juel NG, Liavaag S. Patellofemoral pain: One year results of a randomized trial comparing hip exercise, knee exercise, or free activity. Scand J Med Sci Sports. 2020 Apr;30(4):741-753. doi: 10.1111/sms.13613. Epub 2020 Jan 5. PMID 31846113
- [Background] Constantinou A, Mamais I, Papathanasiou G, Lamnisos D, Stasinopoulos D. Comparing hip and knee focused exercises versus hip and knee focused exercises with the use of blood flow restriction training in adults with patellofemoral pain. Eur J Phys Rehabil Med. 2022 Apr;58(2):225-235. doi: 10.23736/S1973-9087.22.06691-6. Epub 2022 Jan 5. PMID 34985237